CLINICAL TRIAL: NCT01489501
Title: Multicenter Study of Cultured Autologous Oral Mucosal Epithelial Cell-Sheet (CAOMECS) Transplantation to Patients With Total Limbal Stem Cell Deficiency
Brief Title: Multicenter Study of CAOMECS Transplantation to Patients With Total Limbal Stem Cell Deficiency
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Change of strategic priorities in the sponsor's clinical development sector.
Sponsor: CellSeed France S.A.R.L. (Industry)
Collaborators: FGK Clinical Research GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CS001-EU01; 2011-000598-30 (EudraCT Number)
Record Dates: First submitted 2011-12-08; First posted 2011-12-09 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2015-03

CONDITIONS: Limbal Stem Cell Deficiency
Keywords: Caomecs, Transplantation, Limbal stem cell deficiency,
MeSH Terms: conditions — Limbal Stem Cell Deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- only one arm available (Experimental): Caomecs transplantation on eye cornea.
  Interventions: Procedure: Surgical transplantation of CAOMECS to the ocular surface

INTERVENTIONS:
Procedure: Surgical transplantation of CAOMECS to the ocular surface — Surgical transplantation of oral mucosa derived CAOMECS sheet onto eye cornea.

SUMMARY:
This clinical study is a scientific study on patients who do not have any limbal stem cells. In this clinical study tissue is taken from the inside of the mouth, and cells from that tissue (epithelial cells) will be grown to form a multilayered cell-sheet, called CAOMECS, which is then transplanted onto the cornea. This transplantation method should repair the damage of the cornea.

The aim of this study is to see if the transplantation of CAOMECS renews the surface of the eye, by preventing the growth of the conjunctiva over the cornea and stopping new small blood vessels forming.

DETAILED DESCRIPTION:
This is an open clinical study without a control group, which means that all patients will be given the study treatment (CAOMECS).

Adults as well as minor patients can participate in this clinical trial.

CAOMECS is undergoing a clinical trial, which means that it has not yet been officially approved for the treatment of this disease. Up to now it was clinically tested in France, on 26 people with limbal stem cell loss.

Study objective

The objective of this study is to restore the ocular surface epithelium of patients with total LSCD by preventing or reducing recurrent conjunctivalization and neovascularization up to 12 months post-transplantation.

Methodology

This is a prospective, open, multi-center study with CAOMECS in patients with total LSCD. Stem cells will be isolated from an oral mucosa biopsy and will be grown in cell culture. The resultant epithelial cell-sheets will then be transplanted to the ocular surface of the respective patients under general anesthesia. After transplantation patients may be hospitalized according to routine clinical practice.

Overall, the study will consist of a screening visit where eligibility will be evaluated, the day of the biopsy, the day before the transplantation where baseline data will be evaluated, the transplantation (day 0), and a follow-up period consisting of nine visits at days 1, 5, and 10 and months 1, 3, 6, 12, 24, and 36. Other visits as clinically indicated may also occur.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥2 years to 74 years
2. Males or females with bilateral or unilateral total LSCD due to one of the following causes:

   1. Chemical burns
   2. Thermal burns
   3. Contact lens wear
   4. Surgery of the ocular surface
   5. Stevens-Johnson syndrome and other inflammatory disease under stable condition
   6. Aniridia
3. Documented conjunctivalization of the corneal surface, measured by fluorescein staining
4. Stable disease, i.e. history of LSCD for at least 6 months
5. Clinical signs indicative of conjunctivalisation:

   1. Superficial blood vessels on the corneal surface
   2. Loss of epithelial transparency or persistent epithelial defect
6. Healthy oral mucosa
7. Absence from tobacco and alcohol (7 days before the biopsy)
8. Regular tooth brushing (at least twice daily)
9. Ability to comply with the protocol
10. Covered by a social security system
11. Signed informed consent form, ability to understand the study procedures, and contractual capability. Applicable to patient or legal carer (including parent)

    Special inclusion criteria for patients between 18 and 74 years of age (adults):
12. Multiple surgeries in the limbal region

Exclusion Criteria:

1. Acute systemic infection
2. Acute ocular inflammation in the previous 6 months
3. Previous neoplastic/cancer disease
4. Severe dry eye confirmed by a Schirmer test
5. Lyell-Syndrome, epidermolysis bullosa
6. Total symblepharon
7. Medical history of hypersensitivity or allergy to bovine or murine derived materials
8. Pregnant and lactating patients, positive urine pregnancy test in women of childbearing potential
9. Any systemic infectious disease as diagnosed by serology tests such as syphilis, HIV-1, HIV-2, hepatitis B or C, or HTLV-1 infection at screening and at the day of the biopsy
10. Current or previous (within 30 days of enrolment) treatment with another investigational drug or participation in another clinical study
11. Previous participation of the patient in this study
12. Evidence of any other medical conditions (such as psychiatric illness, physical examination or laboratory findings) that may interfere with the planned treatment, affect patient compliance or place the patient at high risk of treatment-related complications
13. Employees of the sponsor or patients who are employees or relatives of the investigator
14. Genetic conditions such as ectodermal dysplasia or multiple endocrine neoplasia

    Special exclusion criteria for patients ≥2 and <18 years of age (children):
15. Multiple surgeries in the limbal region

Ages: 2 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Presence of a stable epithelium on cornea and absence of conjunctivalization in the visual axis | month 12
  This is assessed by delayed fluorescein staining and impression cytology.
Extent of neovascularization | month 12
  Measurement of the area of corneal neovascularisation as documented by photographs.

SECONDARY OUTCOMES:
Presence of a stable epithelium on cornea and absence of conjunctivalization in the visual axis | month 24 and 36
  This is assessed by delayed fluorescein staining and impression cytology.
Extent of neovascularization | month 24 and 36
  Measurement of the area of corneal neovascularisation as documented by photographs.

CONTACTS AND LOCATIONS:
Overall Officials: Friedrich Kruse, Prof. Dr., Principal Investigator — Medizinische Fakultät der Friedrich-Alexander-Universität Erlangen-Nürnberg
Locations (1):
- Universitätsklinkum Erlangen, Erlangen, Bavaria, Germany